CLINICAL TRIAL: NCT00222690
Title: Living With Fibromyalgia (FM): Triggers,Clinical Subgroups, and the Effects Of A Self-Monitored Cognitive-Behavioral and Interactive Technology-Based Intervention on Clinical Subgroups
Brief Title: Living With Fibromyalgia: Triggers,Subgroups, and a Cognitive-Behavioral and Interactive Technology-Based Intervention
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: SHRS Research Development Fund (Unknown); U.S. Department of Education (U.S. Federal Agency)
Other Study IDs: 0505178
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2005-09

CONDITIONS: Fibromyalgia
Keywords: qualitative interview; symptom triggers; activity and participation
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of this study is to conduct semi-structured qualitative interviews to examine the personal experiences of women living with fibromyalgia. The specific aims of this study are to identify clinically relevant "triggers" of fibromyalgia symptoms and examine their impact on activity limitations and participation restrictions.

DETAILED DESCRIPTION:
Fibromyalgia (FM) may currently be the most common rheumatic diagnosis of rheumatologists among their female patients, with 15-20% of all new rheumatology referrals meeting the 1990 American College of Rheumatology (ACR) diagnosis criteria for fibromyalgia. People with fibromyalgia live through widespread musculoskeletal chronic pain, fatigue, psychological distress, and exhibit diminished physical performance due in part to the cycle of pain that adversely affect their activity participation and overall well-being.

The purpose of this prospective mixed methods study is to conduct semi-structured qualitative interviews using ethnographic techniques to examine the personal experiences of women living with fibromyalgia. The specific aims of this study are to identify clinically relevant "triggers" of fibromyalgia symptoms and examine their impact on activity limitations and participation restrictions.

ELIGIBILITY:
Inclusion Criteria:

(1)At least 18 years of age; (2) meet the American College of Rheumatology (ACR) criteria for FM as diagnosed by a physician; (3) have been diagnosed with FM at least 1 year prior to admission to the study; (4) have sufficient vision, based on a functional vision test (i.e., read newsprint) to operate a computer program; (5) speak English; and (6) have a private telephone line.

Exclusion Criteria:

(1)Living beyond a 40-mile radius from the Oakland campus of the University of Pittsburgh. (2)Disability in everyday tasks related to a diagnosis other than FM (e.g., stroke, Parkinson disease) will also be grounds for exclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Hazel L Breland, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh - Department of Occupational Therapy, Pittsburgh, Pennsylvania, United States